CLINICAL TRIAL: NCT00689819
Title: Pre-clinical Cardiac Dysfunction Among Asymptomatic Hypertensive Patients in an Urban Emergency Department: Is a Program Focused on Early Detection and Blood Pressure Control Clinically and Cost Effective?
Brief Title: Pre-clinical Cardiac Dysfunction Among Asymptomatic Hypertensive Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Phillip D. Levy, Research Investigator, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0803305872
Record Dates: First submitted 2008-06-02; First posted 2008-06-04 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-11

CONDITIONS: Hypertension; High Blood Pressure; Ventricular Hypertrophy; Diastolic Dysfunction; Systolic Dysfunction
Keywords: Hypertension; High blood pressure; Pre-clinical cardiac dysfunction
MeSH Terms: conditions — Hypertension | interventions — Exercise; Diet, Sodium-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BP < 140/90 mmHg (Active Comparator): This arm will target a blood pressure of < 140/90 mmHg (or < 130/90 mmHg for diabetics or those with chronic kidney disease) as indicated by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure.
  Interventions: Behavioral: Exercise; Behavioral: Weight Loss; Behavioral: Low Sodium Diet; Behavioral: Smoking Cessation; Drug: Pharmaceutical Therapy (no specific therapy; approach guided by the JNC 7 protocol guidelines)
- BP < 120/80 mmHg (Experimental): This arm will target a more aggressive blood pressure target of < 120/80 mmHg.
  Interventions: Behavioral: Exercise; Behavioral: Weight Loss; Behavioral: Low Sodium Diet; Behavioral: Smoking Cessation; Drug: Pharmaceutical Therapy (no specific therapy; approach guided by the JNC 7 protocol guidelines)

INTERVENTIONS:
Behavioral: Exercise — Blood pressure (BP) target of < 140/90 mmHg (or < 130/80 mmHg for diabetics or with chronic kidney disease) as recommended by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure (JNC 7). BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 140/90 mmHg
Behavioral: Exercise — Blood pressure (BP) target will be < 120/80 mmHg. BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 120/80 mmHg
Behavioral: Weight Loss — Blood pressure (BP) target of < 140/90 mmHg (or < 130/80 mmHg for diabetics or with chronic kidney disease) as recommended by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure (JNC 7). BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 140/90 mmHg
Behavioral: Low Sodium Diet — Blood pressure (BP) target of < 140/90 mmHg (or < 130/80 mmHg for diabetics or with chronic kidney disease) as recommended by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure (JNC 7). BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 140/90 mmHg
Behavioral: Smoking Cessation — Blood pressure (BP) target of < 140/90 mmHg (or < 130/80 mmHg for diabetics or with chronic kidney disease) as recommended by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure (JNC 7). BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 140/90 mmHg
Drug: Pharmaceutical Therapy (no specific therapy; approach guided by the JNC 7 protocol guidelines) — Blood pressure (BP) target of < 140/90 mmHg (or < 130/80 mmHg for diabetics or with chronic kidney disease) as recommended by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure (JNC 7). BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 140/90 mmHg
Behavioral: Weight Loss — Blood pressure (BP) target will be < 120/80 mmHg. BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 120/80 mmHg
Behavioral: Low Sodium Diet — Blood pressure (BP) target will be < 120/80 mmHg. BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 120/80 mmHg
Behavioral: Smoking Cessation — Blood pressure (BP) target will be < 120/80 mmHg. BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 120/80 mmHg
Drug: Pharmaceutical Therapy (no specific therapy; approach guided by the JNC 7 protocol guidelines) — Blood pressure (BP) target will be < 120/80 mmHg. BP control efforts will be open-label and will include a combination of recommended life-style modifications (i.e., exercise, weight loss, low sodium diet, smoking cessation), and pharmaceutical therapy based on JNC 7 protocol driven guidelines with the following adaptations: 1) use of a diuretic that is appropriate to renal function (eGFR< 40 ml/min/1.73 m2: a loop diuretic; eGFR> 40 ml/min/1.73 m2: a thiazide); 2) use of automated reminders if BP exceeds target for > 4 weeks without a medication titration; 3) use of a second diuretic when taking 4 or more anti-hypertensives without adequate achievement of BP target level; and 4) automated alerts to study personnel for potential drug interactions.
  Arms: BP < 120/80 mmHg

SUMMARY:
This project will evaluate the clinical and cost effectiveness of a novel, multidisciplinary approach to identify and treat pre-clinical cardiac dysfunction (PCCD) in asymptomatic hypertensive patients identified in a single center urban emergency department. Premature onset of pressure-related cardiac complications of hypertension (especially heart failure) has important implications for long-term survival, quality of life and healthcare costs. This project will target patients who have already developed pressure-related cardiac structural abnormalities yet remain symptom free. These individuals are at tremendous risk for progression to clinically overt heart failure and its associated consequences. We hypothesize that detection and treatment of patients with hypertension who have pre-clinical structural cardiac damage will enable forestallment of the disease process and offer the opportunity to reduce the burden of cardiac morbidity associated with hypertension. This project will implement a program to prospectively identify PCCD (using echocardiography) and provide treatment. At present, the optimal blood pressure goal for patients with PCCD is unknown so this study will randomize patients to 2 levels of blood pressure control: "normal", which is consistent with current national guidelines and "intensive", which will aim for a markedly lower blood pressure (< 120/80). Enrolled patients will receive active treatment and follow-up for 1 year. At the end of 1 year, we will evaluate: 1) the ability of this program to achieve blood pressure goals; 2) the cost effectiveness; and 3) the proportion in each blood pressure group who have evidence of disease regression on echocardiography.

ELIGIBILITY:
Inclusion Criteria:

* Blood pressure > or = 140/90 after 1 hour
* Asymptomatic state as defined by Goldman Specific Activity Scale

Exclusion Criteria:

* Dyspnea (exertional or nocturnal) or chest pain as a primary or secondary chief complaint
* Prior history of heart failure, coronary artery disease, myocardial infarction, cardiomyopathy, valvular heart disease or renal failure (with current, previous, or planned future dialysis)
* Patients with acute illness or injury which necessitates hospital admission
* Standing relationship with usual source of health care (i.e., primary care provider)

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2008-10; Primary Completion 2011-05 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Phillip D. Levy, M.D., M.P.H., Principal Investigator — Wayne State University Department of Emergency Medicine
Locations (1):
- Detroit Receiving Hospital, Detroit, Michigan, United States

REFERENCES:
- [Derived] Levy PD, Burla MJ, Twiner MJ, Marinica AL, Mahn JJ, Reed B, Brody A, Ehrman R, Brodsky A, Zhang Y, Nasser SA, Flack JM. Effect of Lower Blood Pressure Goals on Left Ventricular Structure and Function in Patients With Subclinical Hypertensive Heart Disease. Am J Hypertens. 2020 Sep 10;33(9):837-845. doi: 10.1093/ajh/hpaa108. PMID 32622346

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment 1: This arm will target a blood pressure of < 140/90 mmHg (or < 130/90 mmHg for diabetics or those with chronic kidney disease) as indicated by the 7th Joint National Committee on Prevention, Detection, Evaluation and Treatment of High Blood Pressure.
- Treatment 2: This arm will target a more aggressive blood pressure target of < 120/80 mmHg.
Period: Overall Study
Arm/Group | Treatment 1 | Treatment 2
Started | 65 | 58
Completed | 45 | 43
Not Completed | 20 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment 1 | Treatment 2 | Total
Number analyzed (Participants) | 65 | 58 | 123
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 65 | 58 | 123
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.3 (8.1) | 49.6 (8.3) | 49.4 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 36 | 80
  Male | 21 | 22 | 43
Region of Enrollment [Number; unit: participants]
  United States | 65 | 58 | 123

OUTCOME MEASURES:

1. Primary Outcome: Clinically Significant Difference in Blood Pressure Lowering, Health Status and Quality of Life
Description: To evaluate the ability of this program to produce (as a surrogate for heart failure prevention) a clinically significant difference in blood pressure lowering, health status and quality of life between the 2 treatment groups.
Time Frame: Baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: mm Hg
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 45 | 43
mm Hg | -3.3 [-7.6 to 2.1] | -4.9 [-11.7 to 1.9]

2. Secondary Outcome: Change in Prevalence of PCCD
Description: To measure the change from baseline to 1 year prevalence of pre-clinical cardiac dysfunction in randomized study patients.
Time Frame: Baseline and 1 year
Measure: Number; unit: percentage of participants
Arm/Group | Treatment 1 | Treatment 2
Number analyzed (Participants) | 45 | 43
percentage of participants | 91.8 | 88.7

ADVERSE EVENTS:
Arm/Group | Treatment 1 | Treatment 2
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/58
Other Adverse Events (participants affected / at risk) | 0/65 | 0/58

LIMITATIONS AND CAVEATS:
Despite our best efforts, study retention was hindered by a higher than expected drop-out rate (26.0% overall; 27.7% control and 24.1% intervention).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No